CLINICAL TRIAL: NCT01509833
Title: Efficacy of Low Dose hCG on Oocyte Maturity for Ovarian Stimulation in Poor Responder Women Undergoing ICSI: a Prospective Randomized Controlled Trial
Brief Title: Efficacy of Low Dose hCG on Oocyte Maturity in Poor Responder Women Undergoing Intracytoplasmic Sperm Injection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Royan Institute (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Royan-Emb-013
Record Dates: First submitted 2012-01-05; First posted 2012-01-13 (Estimated); Last update posted 2012-01-13 (Estimated); Status verified 2009-08

CONDITIONS: Infertility
Keywords: ICSI Ovarian stimulation; hCG low dose; Oocyte maturity; poor respond
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- rFSH (Experimental): Administration of recombinant FSH for ovarian stimulation.
  Interventions: Drug: rFSH
- hCG(100IU) (Experimental): Administration of late follicular low dose hCG(100U) for ovarian stimulation.
  Interventions: Drug: hCG
- hCG(200IU) (Experimental): Administration of late follicular low dose hCG(200IU) for ovarian stimulation.
  Interventions: Drug: hCG

INTERVENTIONS:
Drug: rFSH — Administration of rFSH for ovarian stimulation.
  Arms: rFSH
Drug: hCG — Administration of late follicular low dose hCG(100IU) for ovarian stimulation.
  Arms: hCG(100IU)
Drug: hCG — Administration of late follicular low dose hCG(200IU) for ovarian stimulation.
  Arms: hCG(200IU)

SUMMARY:
This study is a prospective, randomized, parallel, controlled trial to assess the efficacy of the late follicular phase administration of low dose hCG on oocyte maturity for ovarian stimulation in 73 poor respond patients undergoing intracytoplasmic sperm injection (ICSI) treatment.

DETAILED DESCRIPTION:
In this study all eligible patients were randomly allocated into three study groups by a permuted block randomization method: group A (control group) received only recombinant FSH, group B received rFSH supplemented by 100IU hCG in the late follicular phase. Group C received rFSH supplemented by 200IU hCG in the late follicular phase.

All of the patients underwent a standard long protocol and received GnRH-a (Suprefact), 0.5cc subcutaneous, started from the day 17 of the preceding cycle and ovulation induction was started 14 days thereafter.

Patients were categorized according to the following stimulation protocols:

Group A (control group): which 300 IU r-FSH was administered for the first 5 days of the stimulation cycle. Then the first ultrasound scan was performed to monitor response. At this stage the dose of rFSH adjusted according to the ovarian response and continued until the day of ovulatory hCG administration.

Group B: rFSH supplemented with daily administration of 100 IU hCG in the late follicular phase based on the follicle size (14mm).

Group C: rFSH supplemented with daily administration of 200 IU hCG in the late follicular phase based on the follicle size (14mm).

To assess the pregnancy outcomes, serum hCG was measured 2 weeks after embryo transfer. Clinical pregnancy was defined by the observation of sac with fetal heart rate on ultrasonography 4 weeks after embryo transfer.

ELIGIBILITY:
Inclusion Criteria:

1. Poor ovarian response to ovulation induction according to the ESHRE definition[20] and presence of at least 2 of the criteria needed to define poor responders including advanced maternal age, history of low ovarian response in previous IVF/ICSI treatments and abnormal ovarian reserve test(Antral Follicle number < 5)
2. indication for ICSI treatment, second or third cycle
3. Age 37 to 43 years
4. Body mass index (BMI) ≤ 30 kg/m2
5. The presence of two functional ovaries and no previous ovarian surgery
6. The presence of normal uterine cavity and 2 normal tubes base on recent hysterosalpingographic or hysteroscopic evaluation
7. Basal (day 2 or 3) serum FSH levels ≤13 IU/L
8. Normal semen analysis
9. No history or signs of endometriosis
10. No untreated endocrinologic disease

Ages: 37 Years to 43 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2009-10; Primary Completion 2011-03 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Number of mature oocytes | Up to 2 hours after oocyte retrieval
  Evaluation the number of mature oocytes Up to 2 hours after oocyte retrieval

SECONDARY OUTCOMES:
Number of retrieved oocytes | Up to 1 hour after oocyte retrieval
  Evaluation the number of retrieved oocytes Up to 1 hour after oocyte retrieval
Number of generated embryos | Up to 48-72 hours after oocyte retrieval
  Evaluation the number of generated embryos up to 48-72 hours after oocyte retrieval.
Quality of generated embryos | Up to 48-72 hours after oocyte retrieval
  Evaluation the Quality of generated embryos up to 48-72 hours after oocyte retrieval.
Number of transferred embryos | on the time of embryo transfer
  Evaluation the number of transferred embryos on the time of embryo transfer.
Quality of transferred embryos | on the time of embryo transfer
  Evaluation the quality of transferred embryos on the time of embryo transfer.
implantation rate | 4 weeks after embryo transfer
  Evaluation the implantation rate 4 weeks after embryo transfer.
chemical pregnancy rates | 2 weeks after embryo transfer
  Evaluation the chemical pregnancy rates 2 weeks after embryo transfer.
clinical pregnancy rates | 4 weeks after embryo transfer
  Evaluation the clinical pregnancy rates 4 weeks after embryo transfer.

CONTACTS AND LOCATIONS:
Overall Officials: Hamid Gourabi, PhD, Study Chair — Head of Royan Institute; Tahereh Madani, MD, Study Director — scientist; Ladan Mohmmadi yeganeh, MSc, Principal Investigator — scientist
Locations (1):
- Royan Institute, Tehran, Iran

REFERENCES:
- [Derived] Madani T, Mohammadi Yeganeh L, Khodabakhshi S, Akhoond MR, Hasani F. Efficacy of low dose hCG on oocyte maturity for ovarian stimulation in poor responder women undergoing intracytoplasmic sperm injection cycle: a randomized controlled trial. J Assist Reprod Genet. 2012 Nov;29(11):1213-20. doi: 10.1007/s10815-012-9854-3. Epub 2012 Sep 7. PMID 22956348